CLINICAL TRIAL: NCT03839043
Title: Perioperative Smoking Cessation in Surgical Patients Using Short Messaging Service Program.
Brief Title: Short Messaging Service Program to Help Quit Smoking During Perioperative Period.
Acronym: SMS2QUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David Warner, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-010950
Record Dates: First submitted 2019-02-05; First posted 2019-02-15 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Tobacco Use Cessation; Perioperative/Postoperative Complications; Tobacco Smoking
Keywords: Tobacco; Cigarettes; Surgery; Text Message; SMS
MeSH Terms: conditions — Tobacco Use Cessation; Postoperative Complications; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Two hypotheses will be tested using a randomized controlled trial of 200 cigarette smokers scheduled for elective surgery that are willing to maintain temporary abstinence from cigarettes. Using a validated decision aid, subjects stratify according to intended duration of abstinence and randomize within each stratum to receive either a "quit for a bit" or a "quit for good" intervention. Both stratums employ a Short Message Service (SMS or "text") to deliver extended follow-up and assess engagement, e.g. subject response to text requests (ex. # of cigarettes smoked). The "quit for a bit" intervention targets abstinence in the first 7 days after surgery, and has an option of receiving continued messages. Both interventions can continue messages beyond day 30. We will assess treatment engagement outcomes and the continuation rate. We will also obtain biochemically-confirmed abstinence data on the morning of surgery and 30 days post-surgery, as well as self-reported abstinence.
Who Masked: Participant
Masking Description: A randomization schedule for each strata will be generated by the biostatistician using variable length blocks of size 2 or 4 to ensure that the number of subjects assigned to each of the 2 intervention groups remains balanced within each strata. Using these randomization schedules, a computer application program will be used that allows the study personnel to enroll a patient into the trial and obtain the appropriate treatment assignment. The computer application will assign this patient the next sequential treatment assignment for the admission status, and update the randomization dataset accordingly.Once treatment assignment is determined, study personnel will deliver the assigned intervention. The patient will be blinded to treatment assignment to the extent of not knowing the goal of the intervention a priori.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Quit for a bit" (Experimental): Brief behavioral intervention (~5 min) that focus on quitting smoking from the morning of surgery until one week after surgery + "Quit for a bit" SMS program.
  Interventions: Behavioral: Brief behavioral intervention; Other: SMS Program
- "Quit for good" (Active Comparator): Brief behavioral intervention (~5 min) that focus on quitting smoking permanently for as long as possible +" Quit for good" SMS program.
  Interventions: Behavioral: Brief behavioral intervention; Other: SMS Program

INTERVENTIONS:
Behavioral: Brief behavioral intervention — "Quit for a bit"- *advice to quit from the am. of surgery until one week post-surgery, a special emphasis on morning abstinence* risks of smoking to perioperative outcomes, includes wound infections, breathing problems, and heart problems*reduction of these risks if able to quit for a bit*the fact that most smokers don't experience cravings or increased stress around the time of surgery. Subjects will receive written summarizing instructions and a brief abstinence brochure. "Quit for good"- 3 out of the 5A's smoking cessation intervention, including Asking, Advising and Assistance will be provided. The advice endorses immediate, sustained quitting (quit for good), accent on the health and economic benefits of long-term abstinence. Assistance includes a method of setting the date of surgery as the quit date, enlisting social support, anticipation of withdrawal symptoms, and the need for complete abstinence. Subjects will receive written summarizing instructions and a 5As brochure.
Other: SMS Program — "Quit for a bit"- Subjects will get SMS messages focused on maintaining abstinence from the morning of surgery until one week after surgery. SMS content focus on the benefits of abstinence to surgical recovery rather than sustained benefits to overall health. Around day 7 postoperatively, messages will encourage subjects to consider extending their abstinence beyond 7 days."Quit for good"- Subjects will get SMS messages focused on general advice for maintaining abstinence, focusing on the long-term health benefits rather immediate benefits to recovery from surgery. SMS content focus on the the surgical date as the quit date, general advice and support for quitting based on the standard Truth Initiative (UbiQUITxt) message library and there will be no references to effects of short-term abstinence on surgical outcomes.

SUMMARY:
Smoking can increase the risk of complications around the time of surgery. Researchers are trying to see if a text messaging program can help smokers stay off cigarettes around the time of surgery.

DETAILED DESCRIPTION:
The long-term goal of the project is to increase the reach and effectiveness of tobacco use interventions in healthcare settings. The main objective of this project is to determine whether an innovative tobacco use intervention targeting abstinence from the morning of surgery until one week after surgery ("quit for a bit") can increase sustained engagement of surgical patients in treatment compared with a standard tobacco use intervention that specifically targets long-term abstinence ("quit for good").

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Greater than 100 cigarettes lifetime consumption and history of smoking cigarettes every day or most days within the week prior to enrollment
* Willingness to either "quit for a bit" or "quit for good" in the perioperative period, and;
* Owning a device with access to SMS with an unlimited text plan

Exclusion Criteria:

* Surgery on the day of POE evaluation
* Any active psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who elect to continue participating in the SMS service after postoperative day 30 | 30 days Post Op
  Provides one measure of subject engagement in treatment - how many are willing to continue using the text messaging service after 30 days.
The rate at which subjects respond to any requests for subject response delivered via SMS and/or use of "keywords" sent via SMS by the subjects | Cumulative from Day 1 to Day 30 Post Op
  Another measure of treatment engagement, describing willingness of the subjects to interact with the SMS service

CONTACTS AND LOCATIONS:
Overall Officials: David O Warner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Jose T, Cha S, Graham AL, Amato MS, Schroeder DR, Warner DO. Effect of Messaging Content on Engagement With a Short Messaging Service for Perioperative Smoking Cessation. Nicotine Tob Res. 2023 Jul 14;25(8):1465-1473. doi: 10.1093/ntr/ntad061. PMID 37058426
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials